CLINICAL TRIAL: NCT01189669
Title: Long Chain (LC) n-3 Polyunsaturated Fatty Acids (PUFA) Supplementation in Young Women With Polycystic Ovary Syndrome (PCOS): A Cross-over, Placebo Controlled Dietary Intervention Study
Brief Title: n-3 Polyunsaturated Fatty Acids (PUFA) Supplementation in Young Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Adelaide and Meath Hospital (Other)
Collaborators: University College Dublin (Other)
Responsible Party: Dr James Gibney, The Adelaide and Meath Hospital Incorporating the National Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DDC-UCD-PCOS
Record Dates: First submitted 2010-08-24; First posted 2010-08-27 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2008-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- LC n-3 PUFA (Active Comparator): Supplementation with 4 x 1g fish oil capsules (Seven Seas, Ireland) containing 1.9g combined EPA and DHA daily for 6 weeks.
  Interventions: Dietary Supplement: LC n-3 PUFA (fish oil) Supplement
- Placebo (olive oil) supplement (Placebo Comparator): 4 x 1g olive oil capsules (Millas Inc) were given daily for 6 weeks.
  Interventions: Dietary Supplement: Placebo (olive oil) supplement
- Wash out period (No Intervention): A 6 week wash out period separated the LC n-3 PUFA and the Placebo (olive oil) arms. During this period the subjects took no supplements. This arm was designed to minimise a cross-over effect.

INTERVENTIONS:
Dietary Supplement: LC n-3 PUFA (fish oil) Supplement — 4 x 1g LC n-3 PUFA (fish oil)supplement containing 1.9g EPA and DHA given daily for 6 weeks
  Other Names: LC n-3 PUFA (fish oil); Placebo (PL); Wash-out (WO)
  Arms: LC n-3 PUFA
Dietary Supplement: Placebo (olive oil) supplement — 4 x 1g olive oil capsules were given daily for 6 weeks
  Arms: Placebo (olive oil) supplement

SUMMARY:
This is a dietary intervention study designed to assess the impact of long chain (LC) n-3 polyunsaturated fatty acids (PUFA) in young women with polycystic ovary syndrome (PCOS). Considering that LC n-3 PUFA have been reported to have a beneficial affect on many of the adverse metabolic and hormonal aspects of PCOS, it was hypothesised that dietary supplementation with LC n-3 PUFA would have a beneficial therapeutic impact.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a chronic condition affecting young women of reproductive age. Long-term, safe and efficacious treatments are needed for women with this condition, and dietary therapy may have an important role in its treatment. LC n-3 PUFA have been shown to be potent biological regulators, involved in the amelioration of many of the adverse metabolic risk factors which are often present in women with PCOS. The aim of this study was to explore the impact of LC n-3 PUFA on fasting and post-prandial lipid metabolism, as well as on the hormonal profile of women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Had a positive diagnosis of PCOS as defined according to the NIH criteria as chronic oligomenorrhoea (< 9 menstrual cycles per year) and clinical and/or biochemical evidence of hyperandrogenism, in the absence of other disorders causing the same phenotype. Clinical criteria included hirsutism with a Ferriman-Galwey score greater than 9, acne or male pattern alopecia; biochemical criteria included total-testosterone, androstenedione or dehydroepiandrosterone sulphate (DHEAS) greater than the laboratory reference range.
* Were between the ages of 18 and 40

Exclusion Criteria:

* Were under 18 years or greater than 40 years old,
* Were non-Caucasian
* Were pregnant, lactating or trying to conceive
* Had a body mass index (BMI) <18kg/m2 or >50kg/m2
* Had a recent illness or any chronic illness likely to influence results
* Were taking any medications likely to influence the results including hormonal contraception, antihypertensives, lipid lowering medications, antiplatelet agents, anti-inflammatory agents
* Were taking nutritional supplements
* Consumed greater than 2 portions of oily fish per week

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Fasting lipid metabolism | Following supplementation with LCn-3 PUFA or placebo for 6 weeks

SECONDARY OUTCOMES:
Plasma hormonal profile | Following supplementation with LCn-3PUFA or placebo for 6 weeks
Postprandial lipid metabolism | Following supplementation with LCn-3 PUFA or placebo for 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Gibney, Dr, Principal Investigator — The Adelaide and Meath Hospital, incorporating The National Children's Hospital; Helen M Roche, Prof, Principal Investigator — UCD
Locations (2):
- Ireland (2):
  - Diabetes Day Centre, The Adelaide and Meath Hospital, Dublin, Dublin
  - Nutrigenomics Research Group, UCD, Dublin, Dublin

REFERENCES:
- [Derived] Phelan N, O'Connor A, Kyaw Tun T, Correia N, Boran G, Roche HM, Gibney J. Hormonal and metabolic effects of polyunsaturated fatty acids in young women with polycystic ovary syndrome: results from a cross-sectional analysis and a randomized, placebo-controlled, crossover trial. Am J Clin Nutr. 2011 Mar;93(3):652-62. doi: 10.3945/ajcn.110.005538. Epub 2011 Jan 26. PMID 21270384